CLINICAL TRIAL: NCT05869084
Title: Assessment of Bronchial Obstruction in Adolescents With HIV
Acronym: ResppedHIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP211566; IDRCB: 2021-A02635-36 (Registry Identifier: French Health Authority)
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: HIV
Keywords: antiretrovirals
MeSH Terms: interventions — Respiratory Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pulmonary function tests (Experimental)
  Interventions: Diagnostic Test: pulmonary function tests

INTERVENTIONS:
Diagnostic Test: pulmonary function tests — pulmonary function tests

SUMMARY:
In children, data from the literature find a higher prevalence of asthma in the population treated for HIV. Bronchial hyperreactivity, indicative of chronic inflammation and bronchial obstruction, is also present.

Screening for early peripheral obstruction could therefore make it possible to initiate appropriate anti-inflammatory treatment, if necessary, and early preventive management.

DETAILED DESCRIPTION:
In adults chronically infected with HIV, there is an increased prevalence impaired respiratory function, with a greater occurrence of COPD than in the uninfected population. In children, data from the literature find a prevalence of greater atopy in the HIV-infected pediatric population. Furthermore, a bronchial hyperreactivity or even peripheral bronchial obstruction, indicative of a local chronic inflammation has been found in young adolescents treated since the birth for HIV infection in utero. Screening for early peripheral obstruction in HIV-infected adolescents could therefore make it possible to initiate, if necessary, a anti-inflammatory treatment, and early management to prevent the occurrence of impaired respiratory function in adulthood For this this single-center prospective study chose to perform respiratory function explorations with forced oscillometry with the Endpoint main factor of the peripheral obstruction the R5HZ parameter expressed in % predicted. Patients from 11 to 25 years to whom it was proposed added to that to answer a questionnaire of respiratory quality of life

ELIGIBILITY:
Inclusion Criteria:

* Children over 11 and Under 25-year-old infected with HIV and on antiretrovirals and followed up at Robert Debré hospital for this pathology
* Consent of the holders of parental authority and Patients informed and not objecting to participate in research Exclusion Criteria : •
* Age ≤ 11 years old
* Not treated for HIV
* Patients under guardianship / curatorship

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Resistance measured by forced oscillometry (5hZ) | 24 hours
  Resistance measured by forced oscillometry (5hZ)

CONTACTS AND LOCATIONS:
Overall Officials: Veronique HOUDOUIN, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided